CLINICAL TRIAL: NCT01330186
Title: 18F-FMISO-PET, 18F-FDG-PET/CT, DWI-MRI and DCE-MRI Scans as Predictors of Response to Radiotherapy +/- Chemotherapy in Patients With Anal Cancer.
Brief Title: Predictive Value of FMISO-PET, FDG-PET-CT, DWI-MRI and DCE-MRI Scans for Patients With Anal Cancer Receiving Radiotherapy +/- Chemotherapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Eva Serup-Hansen, MD, Department of Oncology, Herlev Hospital
Other Study IDs: GI 1026
Record Dates: First submitted 2011-04-05; First posted 2011-04-06 (Estimated); Last update posted 2011-04-12 (Estimated); Status verified 2011-04

CONDITIONS: Anal Cancer
MeSH Terms: conditions — Anus Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Anal cancer
  Interventions: Other: FMISO-PET, FDG-PET-CT and Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Other: FMISO-PET, FDG-PET-CT and Magnetic Resonance Imaging (MRI) — This study involves 6 imaging sessions. One FMISO-PET before radiation therapy, one FDG-PET-CT before radiation therapy and one FDG-PET-CT during radiation therapy and tree Magnetic Resonance imaging (MRI) sessions with one session before radiation therapy, one session during radiation therapy and one sessions post radiation.

SUMMARY:
The purpose of the study is to evaluate the predictive value of 18F-fluoromisonidazol-PET (FMISO-PET), 2-18F-fluoro-2-deoxy-d-glukose-PET-CT (FDG-PET-CT), Diffusion-Weighted Magnetic Resonance Imaging (DWI-MRI) and Dynamic Contrast-Enhanced Magnetic Resonance Imaging (DCE-MRI) for patients with anal cancer receiving radiation therapy +/- chemotherapy (Cisplatin and 5-FU).

DETAILED DESCRIPTION:
The study involves tree MRI sessions, two FDG-PET-CT sessions and one FMISO-PET session. The FMISO-PET session is presently not carried out because of delivery problems. The production of 18F-fluoromisonidazol at The Department of Clinical Physiology and Nuclear Medicine, Copenhagen University Hospital Herlev, Denmark has not jet been approved by the Danish Medicines Agency.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of invasive primary squamous cell carcinoma of the anal canal or perianal region.
* TNM stage T1-4, N0-3, M0-1
* Treatment with curative intent
* Age > 18 years
* Able to provide informed consent

Exclusion Criteria:

* Contraindication to MRI imaging
* Cardiac pacemaker
* Major obesity
* Serious claustrophobia
* Other malignant disease (except non-melanoma skin cancer) in a period of 5 years prior to imaging study
* Poorly regulated diabetes mellitus despite insulin
* Pregnancy
* Breast feeding
* Known allergy to iv contrast agent
* Major psychiatric illness which would prevent participation in the imaging study
* Infectious wounds on the legs
* Unacceptable kidney function
* Major language difficulties which would prevent participation in the imaging study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with anal canal or perianal cancer
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-02; Primary Completion 2012-02 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Tumor response | 6-8 weeks post radiation
  * Primary tumor 18-F-deoxyglucose (FDG) uptake before radiation and during week 3 of radiation.
  * Primary tumor apparent diffusion coefficient before radiation and during week 3 of radiation and 6-8 weeks post radiation
  * Primary tumor perfusion coefficient before radiation and during week 3 of radiation and 6-8 weeks post radiation
  * Primary tumor 18-F-Fluoromisonidazol (FMISO) uptake before radiation

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Oncology Herlev Hospital, Herlev, Denmark